CLINICAL TRIAL: NCT04714398
Title: SupportBP 2.0: Behavioral Science and Enrollment in Remote Monitoring for Hypertension Management
Brief Title: SupportBP 2.0:Behavioral Science and Enrollment in Remote Monitoring for Hypertension Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shivan J Mehta, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 844150
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Hypertension
Keywords: blood pressure; remote monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Opt-In Recruitment (Experimental): All recruitment messaging will be framed for patients as they must opt-in to participate in the remote monitoring program.
  Interventions: Behavioral: Opt-In Recruitment
- Opt-Out (Experimental): All recruitment messaging will be framed as though participation is the default, and patients must opt-out of participating in the remote monitoring program.
  Interventions: Behavioral: Opt-Out Recruitment
- Usual Care (No Intervention): Patients in the usual care arm will not be contacted by study staff, they will not receive a blood pressure cuff, and they will not be asked to participate in any component of the blood pressure monitoring program.

INTERVENTIONS:
Behavioral: Opt-In Recruitment — Patients in the opt-in recruitment arm will receive a letter describing the program and inviting them to participate in the remote monitoring program. Along with the letter they will receive an informational brochure and a copy of the informed consent form. Patients in this arm will then receive a recruitment phone call explaining the program and consenting the participant verbally. If the participant consents to participate in the remote monitoring program, to receive text messaging, and to connection to care, the research coordinator will mail a blood pressure cuff and begin the remote monitoring program for the patient 6 days later.
  Arms: Opt-In Recruitment
Behavioral: Opt-Out Recruitment — Patients assigned to opt-out recruitment will receive a blood pressure cuff with instructions in the mail along with a letter describing the program and opt-out framing regarding their participation, as well as a brochure and a copy of the informed consent form. Patients in this arm will receive a recruitment phone call similar to recruitment arm A, explaining the program and consenting the participant verbally. If the participant consents to participate in the remote monitoring program, to receive text messaging, and to connection to care, the research coordinator will begin the remote monitoring program for the patient immediately.
  Arms: Opt-Out

SUMMARY:
A 3-arm randomized pilot trial aimed at comparing the effectiveness of different approaches to recruiting patients to participate in a 6-month remote monitoring program for the management of hypertension (HTN).

DETAILED DESCRIPTION:
The investigators will utilize the Way to Health (WTH) platform to develop and evaluate a new remote monitoring enrollment model that is integrated with routine clinical care at Penn Family Care (PFC), an academic family medicine practice in West Philadelphia. Among patients with poorly controlled HTN the investigators will:

1. Compare the effect of sending eligible patients a blood pressure cuff with the mailed invitation letter and opt-out framing versus the more conventional method of phone calls following mailed letters.
2. Evaluate the feasibility and effectiveness of a remote monitoring program with individualized stepped escalation for hypertension management.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years old with HTN (ICD-10 code I10)
2. Has had at least one office visit at Penn Family Care (PFC) within the past 12 months (at time of chart review), with the last visit having a BP reading exceeding HTN guidelines (150/90 if >60 or, 140/90 if ages 21-59 yrs or has CKD or diabetes).
3. Must have a cellular phone with texting capabilities
4. Must be prescribed at least one medication for hypertension

Exclusion Criteria:

1. Has metastatic (Stage IV) cancer
2. Has end stage renal disease
3. Has congestive heart failure
4. Has dementia
5. BMI >= 50
6. Is Non-English speaking requiring a translator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Proportion Participating by Recruitment Method | 6 months, from date of consent to end of remote monitoring program
  The proportion of patients participating in each study arm out of the number randomized to that study arm.

SECONDARY OUTCOMES:
Proportion Engaged by Recruitment Method | 6 months, from date of consent to end of remote monitoring period
  The proportion of patients recruited by each method who are actively engaged with the program
Proportion with Controlled Blood Pressure by Monitoring vs. Usual Care | 6 months, from date of consent to end of remote monitoring program
  The proportion with controlled blood pressure by remote monitoring and the proportion with controlled blood pressure by clinic visits (usual care).
Blood Pressure Trajectory by Recruitment Method | 6 months, from date of consent to end of remote monitoring program
  The systolic and diastolic blood pressure trajectory by recruitment arm.
Proportion of BP Measurements Submitted by Recruitment Method | 6 months, from date of consent to end of remote monitoring program
  The proportion of requested BP measurements submitted by each patient by recruitment arm

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Teel J, Okorie E, Reitz C, Purcell A, Snider CK, Clark K, Kersting RC, Glanz K, Putt M, Rareshide C, Volpp KG. Behavioral Economic Framing for Enrollment and Retention of Patients in Remote Blood Pressure Monitoring: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2529825. doi: 10.1001/jamanetworkopen.2025.29825. PMID 40892409